CLINICAL TRIAL: NCT07141160
Title: ADL+2.0: Intervention for Prevention of Cognitive Decline in Community-dwelling Older Adults.
Acronym: ADL+ 2
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Nanyang Technological University (Other); Geriatric Education and Research Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ECOS Ref 2024-4524
Record Dates: First submitted 2025-08-04; First posted 2025-08-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Decline
Keywords: Subjective memory complaints; Technology-enabled; Multi-component intervention; Cognitive decline; Intrinsic motivation; Prevention
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This is a type 1 hybrid effectiveness-implementation to ascertain the efficacy, cost-effectiveness, and implementation of the ADL+ 2.0 programme. The effectiveness study will use a cluster randomised trial design that compares 3 participant groups: a) receiving a combination of remote and onsite interventions, b) receiving only remote interventions, and c) education booklet + health talk group.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remote mobile based app (Experimental): Mobile based digital toolkit for cognitive health, remote assessment and multi-component intervention, comprising the 4 key pillars of assessment; cognitive training and stimulation; cognitive wellness; and dual-task training.
  Interventions: Other: Combined: Mobile app + 6WELLS
- Combined: Mobile app + 6WELLS (Experimental): Mobile based digital toolkit for cognitive health, remote assessment and multi-component intervention, comprising the 4 key pillars of assessment; cognitive training and stimulation; cognitive wellness; and dual-task training. Together with onsite 6 WELLS Group-Based Activity is a structured, group-based, cognitive health promotion programme that aims to build communities of practice, stimulate goal attainment, and drive behavioural change towards cognitive health and wellbeing. The curriculum is delivered via a 10-week onsite programme comprising weekly facilitated small-group activities centred on six key components.
  Interventions: Other: Remote mobile based app
- Educational booklet and health talk (Sham Comparator): Education booklet and a health talk on cognition. The booklet and health talk will be provided to the participants, it comprises of tips for maintaining cognitive health. Both aims to promote the awareness for normal ageing and dementia.
  Interventions: Other: Combined: Mobile app + 6WELLS; Other: Remote mobile based app

INTERVENTIONS:
Other: Combined: Mobile app + 6WELLS — Mobile based digital toolkit for cognitive health, remote assessment and multi-component intervention, comprising the 4 key pillars of assessment; cognitive training and stimulation; cognitive wellness; and dual-task training. Together with onsite 6 WELLS Group-Based Activity is a structured, group-based, cognitive health promotion programme that aims to build communities of practice, stimulate goal attainment, and drive behavioural change towards cognitive health and wellbeing. The curriculum is delivered via a 10-week onsite programme comprising weekly facilitated small-group activities centred on six key components.
  Arms: Educational booklet and health talk; Remote mobile based app
Other: Remote mobile based app — Mobile based digital toolkit for cognitive health, remote assessment and multi-component intervention, comprising the 4 key pillars of assessment; cognitive training and stimulation; cognitive wellness; and dual-task training.
  Arms: Combined: Mobile app + 6WELLS; Educational booklet and health talk

SUMMARY:
Singapore's rising dementia incidence with an ageing population presents an urgent need for effective interventions that delay or prevent cognitive decline. While multi-domain intervention studies for dementia prevention show promise, there is a need for an effective personalised approach to address an individual's multifactorial risks for dementia, and to achieve cost-effective, scalable and sustainable outcomes for wider implementation.

The investigators propose the ADL+ 2.0 programme, an overall goal is to delay or prevent cognitive decline in at-risk individuals without dementia aged 60 and above with subjective memory complaints and/or impaired cognitive capacity from the ICOPE screening tool. Through a population-level, technology-enabled, community-based preventative approach, ADL+ 2.0 provides remote assessment and multi-component intervention (cognitive training, dual-task exercises, and cognitive wellness) with smart scheduling and personalized intervention, and can be delivered in conjunction with the onsite 6 WELLS facilitated group-based activity, underpinned by the Self-Determination Theory to foster intrinsic motivation for lasting behavioural change.

The approach begins with phase 1 test-bedding approach Type 1 hybrid effectiveness-implementation study to ascertain the efficacy, cost-effectiveness, and implementation of the ADL+ 2.0 programme. The investigators will conduct a 3-arm cluster-randomised controlled trial comparing remote/onsite, remote only, and control groups to assess the impact on cognitive outcomes, social networks, quality-of-life and cost-effectiveness. Barriers and facilitators will be identified for implementation, guided by the Consolidated Framework for Implementation Research.

Together with NTU-LILY/LKCMedicine as technology partner and community partners (NTUC Health, Fei Yue Community Services, and evaluation partners (GERI/NUS) to provide evidence for and effectively implement a scalable, sustainable, and cost-effective community programme for the prevention of cognitive decline in Singapore.

DETAILED DESCRIPTION:
An estimated one in 10 people aged 60 and above in Singapore suffers from dementia. With increasing life expectancy and a rapidly ageing population, the number of persons living with dementia is expected to continue to rise, with significant negative consequences at individual, societal and healthcare system levels. To address this problem, multidomain non-pharmacological interventions aimed at addressing various risk factors for dementia prevention hold promise. However, a gap exists in overcoming practical barriers, demonstrating cost-effectiveness, and ensuring scalability and sustainability of these interventions.

To address these gaps, the investigators propose ADL+ 2.0: Intervention for prevention of cognitive decline in community-dwelling older adults. The ADL+ 2.0 programme takes a population-level, technology-enabled, community- based preventative approach, targeting community-dwelling individuals without dementia aged 60 years and above who are at risk of cognitive decline. Type 1 hybrid effectiveness-implementation study will be conducted to ascertain the efficacy, cost-effectiveness, and implementation of the ADL+ 2.0 programme.

Firstly, to determining the effectiveness of the ADL+ 2.0 programme in improving cognition, social participation, and health-related quality of life amongst older persons at risk of cognitive decline serves as a pre- requisite before further implementation and scaling in the community. Secondly, determining the cost-effectiveness of the ADL+ 2.0 programme is important to understand the funding and resource implications for longer-term sustainability. Lastly, explicating the facilitators and barriers for participation/adherence at the individual user level and delivery of programme at the systems level will enable the study team to develop implementation strategies and further refine and develop the ADL+ 2.0 intervention in the scale up (deployment) phase.

ELIGIBILITY:
Inclusion Criteria:

* ≥60 Years old
* Participants from partnering Active Ageing Centres (AACs) across Singapore
* Subjective memory complaint (AD8 ≥ 2)
* Independent in activities of daily living (ADL)
* Able to speak English and/or Mandarin
* Comfortable with using smartphones
* Not currently enrolled in a formal cognitive training program.

Exclusion Criteria:

* Known dementia or suspected dementia after initial screening
* Significant medical illnesses

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2029-08-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive test performance | Through study completion, an average of 9 months
  The primary efficacy outcome will be change in cognitive test performance in composite and individual domain z- scores using a standardised neuropsychological test battery (NTB) comprising the 5 domains of attention, processing speed, memory, language, and executive function.

SECONDARY OUTCOMES:
Efficacy outcomes - Cognition | through study completion, an average of 9 month
  The investigators will assess subjective memory complaints using the locally validated AD8 questionnaire. Possible scores range from 0-1 (normal cognition) to 2-8 (cognitive impairment is likely to be present).
Efficacy outcomes - Function & Social | through study completion, an average of 9 month
  Investigators will look at the transfer of cognitive benefits to activities of daily living using the Alzheimer's Disease Cooperative Study- Activities of Daily Living Prevention Instrument (ADCS-PI). The ADCS-PI consists of 15 IADL tasks and 5 physical function questions. Lubben Social Network Scale (LSNS-6) will be used to assesses the domains of social isolation and Frenchay Acitivities Index to assess participation in social activities.
Efficacy outcomes - Quality of Life | through study completion, an average of 9 month
  Health-related quality of life (QOL) will be assess using the 5-level EuroQol 5-dimension (EQ-5D-5L) to derive utility scores based on Singapore preference weights derived using an indirect interim mapping method, and to estimate quality adjusted life years (QALY). 11-item Control, Autonomy, Self-realisation, and Pleasure (CASP-11) tool, which was developed specifically to assess emotional QOL in older adults. CASP-11 has a total score range of 0 to 33. A higher score indicates a higher quality of life.

OTHER OUTCOMES:
Cost analysis evaluation | through study completion, an average of 9 month
  Investigators will conduct a cost-effectiveness analysis based on two efficacy outcomes to determine the incremental cost-effectiveness ratio, namely the neuropsychological test battery (NTB) Z-score, and quality-adjusted life-years to be computed from EQ-5D results. An estimate of the implementation and intervention cost per study participant and cost per site. This will support a comparison of the two intervention arms (remote and onsite, remote only), and inform the study team on the resources required for Phase 2.
IAM (Intervention Appropriateness Measure) score | through study completion, an average of 9 month
  To understand the implementation strategies, qualitative interviews will be conducted to understand the adherence of the ADL+ 2.0. The scale values range from 1 to 5, higher scores indicate greater appropriateness
FIM (Feasibility of Intervention Measure) scale | through study completion, an average of 9 month
  To understand the implementation strategies, qualitative interviews will be conducted to understand the adherence of the ADL+ 2.0 with FIM (Feasibility of Intervention Measure) scale. The scale values range from 1 to 5, higher scores indicate greater feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Wee Shiong Lim, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No